CLINICAL TRIAL: NCT07174583
Title: A Multicenter Study Evaluating the Safety, Efficacy, and Pharmacokinetics of IDE849 in Patients With DLL3-Expressing Tumors Including Small Cell Lung Cancer
Brief Title: A Study of IDE849 in Patients With DLL3 Expressing Tumors Including Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: IDEAYA Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDE849-001
Record Dates: First submitted 2025-09-11; First posted 2025-09-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Small-cell Lung Cancer; Neuroendocrine Carcinomas; Solid Tumor Show to Express DLL3
Keywords: IDE849; Small Cell Lung Cancer; SCLC; anti-DLL3 immunoglobulin G1 monoclonal antibody; DLL3; Neuroendocrine Carcinomas; NEC; durvalumab; IDE161
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Neuroendocrine | interventions — durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Experimental: Part 1A IDE849 Monotherapy (Dose Escalation) (Experimental): Successive cohorts of participants will be treated with escalating doses of IDE849 until the maximum tolerated dose and dose for expansion are determined
  Interventions: Drug: IDE849
- Experimental: Part 1B IDE849 + durvalumab (Dose Escalation) (Experimental): Multiple doses of IDE849 will be tested in combination with durvalumab to identify the optimal combination dose.
  Interventions: Drug: IDE849; Drug: durvalumab
- Experimental: Part 1B IDE849 + IDE161 (Dose Escalation) (Experimental): Multiple doses of IDE849 will be tested in combination with IDE161 to identify the optimal combination dose.
  Interventions: Drug: IDE849; Drug: IDE161
- Experimental: Part 2 IDE849 Monotherapy (Dose Expansion) (Experimental): Chosen monotherapy doses of IDE849 will be tested in additional participants.
  Interventions: Drug: IDE849
- Experimental: Part 2 IDE849 + durvalumab (Dose Expansion) (Experimental): Chose combination dose of IDE849 + durvalumab will be tested in additional participants.
  Interventions: Drug: IDE849; Drug: durvalumab
- Experimental: Part 2 IDE849 + IDE161 (Dose Expansion) (Experimental): Chose combination dose of IDE849 + IDE161 will be testing in additional participants
  Interventions: Drug: IDE849; Drug: IDE161

INTERVENTIONS:
Drug: IDE849 — IV administration
Drug: durvalumab — IV administration
  Other Names: durvalumab Injection [Imfinzi]
  Arms: Experimental: Part 1B IDE849 + durvalumab (Dose Escalation); Experimental: Part 2 IDE849 + durvalumab (Dose Expansion)
Drug: IDE161 — oral administration
  Arms: Experimental: Part 1B IDE849 + IDE161 (Dose Escalation); Experimental: Part 2 IDE849 + IDE161 (Dose Expansion)

SUMMARY:
This is Phase 1/2, multicenter, clinical study to evaluate the safety, efficacy, PK, and immunogenicity of IDE849 in subjects with DLL3-expressing tumors including SCLC.

DETAILED DESCRIPTION:
This multicenter, open-label, Phase 1/2 study is designed to further characterize the safety, tolerability, pharmacokinetics (PK), immunogenicity, and preliminary anti-tumor activity of IDE849, an anti-DLL3 antibody-drug conjugate, alone and in combination with durvalumab or IDE161, in subjects with DLL3-expressing tumors including small-cell lung cancer (SCLC), high-grade neuroendocrine carcinomas (NEC), and other DLL3-positive solid tumors.

Part 1 (Dose Escalation):

Part 1A will evaluate IDE849 monotherapy, and Part 1B will evaluate IDE849 in combination with durvalumab or IDE161. This phase is designed to assess safety and tolerability, identify dose-limiting toxicities (DLTs), and determine the maximum tolerated dose (MTD) and recommended dose for expansion (RDE), in subjects with extensive-stage SCLC, high-grade NEC, or other DLL3-expressing tumors.

Part 2 (Dose Expansion):

Part 2 further will evaluate IDE849 alone or in combination at selected dose levels to characterize safety, PK, immunogenicity, and preliminary anti-tumor activity in defined cohorts of subjects with extensive-stage SCLC, high-grade NEC, or other DLL3-expressing tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Are willing to participate in this clinical study, understand the study procedures, and are able to sign the written ICF.
2. Subjects with histologically or cytologically confirmed extensive-stage SCLC neuroendocrine carcinoma (NEC), and other DLL3+ tumors, are eligible per protocol. Subjects must have radiologically progressed or recurred after previous standard treatment, For SCLC, this includes platinum-based therapy and programmed death-1/programmed death-ligand 1 inhibitors (except for subjects who refuse or are judged by the Investigator to be unsuitable for immunotherapy). No more than 2 lines of previous systemic chemotherapy in any setting and no more than 3 total lines of systemic therapy in the recurrent or metastatic setting will be allowed.
3. Subjects will be required to provide blood/tumor tissue samples for biomarker testing.
4. Have at least 1 measurable lesion according to RECIST version 1.1.
5. Have Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1.
6. Have life expectancy > 3 months.
7. Have adequate bone marrow and organ function.
8. Women of childbearing potential must agree to take highly effective contraceptive measures from signing of consent through 8 months after the last dose of IDE849; men with partners of child-bearing potential must use effective contraception through 5 months after the last dose.

Exclusion Criteria:

1. Have mixed SCLC and nonsmall cell lung cancer histology (SCLC with components of large cell neuroendocrine carcinoma are eligible).
2. Subjects with locally untreated (radiotherapy or surgery) or active central nervous system (CNS) tumor metastasis.
3. Have had other malignancies within 2 years prior to the first dose, except adequately treated carcinoma in situ (cervical, breast, or other), basal cell or squamous cell skin cancer, localized prostate cancer after curative therapy with no recurrence, or papillary thyroid cancer after curative resection; other prior or concurrent malignancies may be eligible with Medical Monitor review and approval.
4. Have uncontrolled tumor-associated pain.
5. Have severe cardiovascular and cerebrovascular disease
6. Have history of clinically significant bleeding within 3 months before the first study dose.
7. Have history of interstitial pneumonitis during previous treatment; current noninfectious pneumonitis requiring steroid therapy; known or suspected interstitial pneumonitis as seen on screening imaging; other moderate to severe lung diseases seriously affecting respiratory function within 3 months before the first dose, including, but not limited to, idiopathic pulmonary fibrosis and organizing pneumonia/obliterative bronchiolitis.
8. Have history of immunodeficiency, with a positive human immunodeficiency virus (HIV) test.
9. Subjects with known or suspected viral hepatitis.
10. Have a history of active tuberculosis within 1 year before enrollment.
11. For participants enrolling to receive the combination with durvalumab, must not have had any prior Grade 2 or higher myocarditis or any other Grade 3 or higher immune-related AE. If the participant has had a prior immune-related AE, must have recovered to < Grade 1
12. For participants enrolling to receive the combination with IDE161, must not have had prior gastrectomy or upper bowel removal or any other gastrointestinal disorder or defect eg, malabsorption disorder such as Crohn's disease or ulcerative colitis, that would interfere with absorption of IDE161
13. Have received chemotherapy within 3 weeks of first dose of IMP; immunotherapy or biologic targeted anti-tumor treatments within 2 weeks before the first dose of IMP; for small molecule treatments within 2 weeks before the first dose of the IMP or within 5 half lives of the drug (whichever is longer); other investigational products within 4 weeks or within 5 half-lives of the drug (whichever is longer) unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study. Participants who received an immunotherapy agent (eg, PD-1/PD-L1 inhibitor) immediately prior to study enrollment must have documented radiologic disease progression as per the Investigator prior to first dose of IMP
14. Administration of any of the following:

    * Strong inhibitors or inducers of CYP3A4
    * Strong inhibitors of CYP2D6
    * Strong inhibitors of P-gp or BCRP
    * Use of drugs with a known risk of QT prolongation
15. For participants enrolling to receive the combination with IDE161:

    * Use of drugs of narrow therapeutic index that are sensitive substrates of MATE2-K, BCRP, and P-gp
    * Use of known moderate and strong CYP3A4/5 inducers and inhibitors is not permitted
    * Administration of PPIs
    * Use of an H2 blocking agent
    * Use of a local antacid
    * Use of drugs with a known risk of QT prolongation
16. Have prior treatment with DLL3 ADC or prior treatment with a topoisomerase I inhibitor including an ADC with a topoisomerase I inhibitor payload.
17. For participants enrolling to receive the combination with durvalumab, have history of prior intolerance to PD-1/PD-L1 inhibitors
18. Have received > 30 Gy of chest radiotherapy within 12 weeks prior to the first dose of the IMP, > 30 Gy of non-chest radiotherapy within 4 weeks prior to the first dose (subjects who have completed radiotherapy for brain metastases within 14 days prior to the first dose can be enrolled and palliative radiotherapy for other sites of ≤ 30 Gy is allowed if completed more than 14 days prior to the first dose).
19. Have undergone major surgery or experienced significant trauma within 4 weeks prior to the first dose.
20. Female subjects who are pregnant, lactating, or planning to become pregnant during the study period to 8 months after the last dose of the IMP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Part 1A: Safety and Tolerability of IDE849 (Monotherapy) | approximately 4 years total study duration
  Incidence of dose-limiting toxicities, incidence and severity AEs and SAEs as measured by CTCAE V5.0.
Part 1B: Safety and Tolerability of IDE849 in Combination with durvalumab or IDE161 | approximately 4 years total study duration
  Incidence of dose-limiting toxicities, incidence and severity AEs and SAEs as measured by CTCAE V5.0.
Part 2: Safety and Tolerability of IDE849 (Monotherapy Dose Expansion) | approximately 4 years total study duration
  Incidence and severity and relationship of AEs and SAEs as measured by CTCAE V5.0
4. Part 2: Safety and Tolerability of IDE849 in Combination with durvalumab or IDE161 (Dose Expansion) | approximately 4 years total study duration
  Incidence and severity and relationship of AEs and SAEs graded as measured by CTCAE V 5.0.
Part 2: Objective Response Rate (ORR) and Investigator Assessment of IDE849 ORR per RECIST 1.1 | approximately 4 years total study duration
  ORR per RECIST v1.1, defined as the proportion of subjects with a Complete Response (CR) or Partial Response (PR) as assessed by the Investigator.
Part 2: Duration of Response (DOR) and Investigator Assessment of IDE849 DOR per RECIST 1.1 | approximately 4 years total study duration
  DOR per RECIST v1.1, defined as the time from the first documented Complete Response (CR) or Partial Response (PR) to disease progression or death, whichever occurs first, as assessed by the Investigator.

SECONDARY OUTCOMES:
Part 1 and Part 2: Disease Control Rate (DCR) and Investigator Assessment of IDE849 DCR per RECIST 1. | approximately 4 years total study duration
Part 2: Progression-Free Survival (PFS) PFS per RECIST1.1 PFS per RECIST1.1. | approximately 4 years total study duration
Part 2: Overall Survival (OS) | approximately 4 years total study duration
  Overall Survival (OS) defined as the time from first dose of IDE849 to death due to any cause
Part 1 and Part 2: Pharmacokinetics (PK) of IDE849 and in combination with durvalumab and IDE161 Blood concentrations and PK parameters. | approximately 4 years total study duration
6. Part 1 and Part 2: Dose-Exposure Response of IDE849 and in combination with durvalumab and IDE161 Relationship between IDE849 dose level and systemic exposure based on plasma concentration data and pharmacokinetic parameters | approximately 4 years total study duration
Part 1 and Part 2: Dose-Exposure Response of IDE849 and in combination with durvalumab and IDE161 Relationship between IDE849 dose level and systemic exposure based on plasma concentration data and pharmacokinetic parameters | approximately 4 years total study duration

CONTACTS AND LOCATIONS:
Locations (39):
- United States (20):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Mayo Clinic Hospital - Florida, Jacksonville, Florida
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - Piedmont Physicians Medical Oncology - Atlanta, Atlanta, Georgia
  - The University of Chicago Medical Center - Duchossois Center for Advanced Medicine, Chicago, Illinois
  - OSF HealthCare Cancer Institute, Peoria, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc. - Fort Wayne North Office, Fort Wayne, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Trinity Health-IHA Medical Group - Hematology Oncology - Ann Arbor Campus, Ann Arbor, Michigan
  - The Cancer and Hematology Centers, Grand Rapids, Michigan
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - Weill Cornell Medicine - Cutaneous Oncology and Melanoma Program, New York, New York
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute - Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center Houston, Texas 77030-4000, Houston, Texas
  - Oncology Consultants, PA - Houston, Houston, Texas
  - Next Oncology Dallas, Irving, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Private Hospital - Southern Oncology Clinical Research Unit (SOCRU), Bedford Park, South Australia
  - Cabrini Hospital - Malvern, Clayton, Victoria
- Brazil (4):
  - Hospital de Câncer de Barretos - Fundação Pio XII, Barretos, São Paulo
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, São Paulo
  - Faculdade de Medicina de Sao Jose do Rio Preto-SP - Hospital de Base, São José do Rio Preto, São Paulo
  - Next Brasil (Rede D'Or), São Paulo, São Paulo
- Canada (2):
  - University Health Network (UHN) - Princess Margaret Cancer Centre (Princess Margaret Hospital), Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyō City, Tokyo-To, Japan
- South Korea (4):
  - National Cancer Center, Gyeonggi-do, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Samsung Medical Center, Seoul, Seoul
  - Severance Hospital - Yonsei Cancer Center, Seoul, Seoul
- Spain (4):
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - South Texas Accelerated Research Therapeutics Madrid - CIOCC - Universitario Sanchinarro, Madrid, Madrid
  - NEXT Madrid -Hospital Universitario Quiron Salud Madrid, Pozuelo de Alarcón, Madrid
  - Hopsital Universitario Virgen Macarena, Seville, Sevilla